CLINICAL TRIAL: NCT01557192
Title: Low Field Magnetic Stimulation in Mood Disorders in Six Visits
Brief Title: Low Field Magnetic Stimulation (LFMS) in Mood Disorders: 6 Treatments
Acronym: LFMS6tx
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: on hold indefinitely due to lack of funding
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Michael Rohan, Imaging Physicist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-P-001097
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Bipolar Depression; Unipolar Depression
Keywords: Depression; Bipolar Depression; LFMS; Electromagnetic Stimulation
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active LFMS treatment (Active Comparator): 20 minute exposure to the LFMS electromagnetic field treatment
  Interventions: Device: Low Field Magnetic Stimulation Device
- Sham LFMS treatment (Placebo Comparator): 20 minute exposure to either the sham (inactive) electromagnetic field treatment
  Interventions: Device: Low Field Magnetic Stimulation Device

INTERVENTIONS:
Device: Low Field Magnetic Stimulation Device — The Low Field Magnetic Stimulation (LFMS) procedure is an application of a series of electromagnetic pulses to the brain lasting twenty minutes. Subjects will be given one 20 minute exposure to either the LFMS or sham electromagnetic field treatment.
  Other Names: LFMS

SUMMARY:
To demonstrate the efficacy of multiple applications of Low Field Magnetic Stimulation (LFMS) as an antidepressant treatment in subjects with mood disorders.

DETAILED DESCRIPTION:
The Low Field Magnetic Stimulation (LFMS) procedure is an application of a series of electromagnetic pulses to the brain lasting twenty minutes. The field and timing parameters of the LFMS pulses, such as pulse timing, duration, frequency, and electric and magnetic field distribution and direction are different from other neurostimulation methods.

The mechanism of action for the antidepressant effects of LFMS is hypothesized to be an effect on dendritic or synaptic activity in the cortex, brought about by low level electrical stimulation applied with particular timing. This is analogous to the synaptic effects of pharmaceutical antidepressants in providing a "boost" to synapses in certain brain regions.

Previous investigations of LFMS included depressed subjects with bipolar disorder. This study will evaluate the antidepressant effects of multiple LFMS treatments in bipolar disorder and major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects MUST be significantly depressed, currently.
2. Subjects must not have serious physical illnesses, neurological diseases or dementias.
3. Subjects will meet DSM-IV criteria for Bipolar Disorder Type I or II, Major Depressive Disorder, Post Traumatic Stress Disorder, or Obsessive Compulsive Disorder, and be currently depressed.
4. Subject must have a Ham-D score > 17, YMRS score < 7 (bipolar subjects only), and a MADRS score > 18.
5. Subjects must be capable of providing informed consent.
6. Subjects must have an established residence and phone.
7. Subjects may be medicated or unmedicated.

Exclusion Criteria:

1. Dangerous or active suicidal ideation.
2. Pregnant or planning on becoming pregnant.
3. Substance abuse (cannot meet DSM criteria for substance abuse, no significant drug abuse within last 3 months, no major polysubstance abuse history, no history of dependence in last year, no drug use within last month).
4. Mixed mood state or rapid cycling.
5. Presence of a pacemaker, neurostimulator, or metal in head or neck.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS)score | at baseline and at week 3
  MADRS scores will be compared between the baseline and week 3, one week after the final treatment.
Change in Positive-Negative Affect Scale (PANAS)score | at baseline and at one and at week 3
  PANAS scores will be compared between the baseline and week 3, one week after the final treatment.

SECONDARY OUTCOMES:
Immediate mood improvement as measured by the difference in post and pre treatment PANAS ratings | at baseline and immediately before and after each treatment, 6 treatments across 2 weeks
  PANAS scores will be assessed at baseline and before and after each treatment. There are six treatments (Monday, Wednesday and Friday for two weeks).
Change in Montgomery-Asberg Depression Rating Scale (MADRS)score | at baseline and at week 4
  MADRS scores will be compared between the baseline and week 4, two weeks after the final treatment.
Change in Positive-Negative Affect Scale (PANAS)score. | at baseline and at one and at week 4
  PANAS scores will be compared between the baseline and week 4, two weeks after the final treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Rohan, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Rohan M, Parow A, Stoll AL, Demopulos C, Friedman S, Dager S, Hennen J, Cohen BM, Renshaw PF. Low-field magnetic stimulation in bipolar depression using an MRI-based stimulator. Am J Psychiatry. 2004 Jan;161(1):93-8. doi: 10.1176/appi.ajp.161.1.93. PMID 14702256
- [Result] Carlezon WA Jr, Rohan ML, Mague SD, Meloni EG, Parsegian A, Cayetano K, Tomasiewicz HC, Rouse ED, Cohen BM, Renshaw PF. Antidepressant-like effects of cranial stimulation within a low-energy magnetic field in rats. Biol Psychiatry. 2005 Mar 15;57(6):571-6. doi: 10.1016/j.biopsych.2004.12.011. PMID 15780843